CLINICAL TRIAL: NCT04932252
Title: A Dose Block-randomized, Double Blinded, Placebo Controlled, Dose-escalation Clinical Trial to Find the Maximal Tolerable Dose and to Evaluate the Safety, Tolerability and Pharmacokinetics After Single and Multiple Oral Doses of A4368 in Healthy Subjects
Brief Title: A Study of A4368 in Healthy Subjects
Acronym: A4368
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autophagy Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS101
Record Dates: First submitted 2021-06-03; First posted 2021-06-21 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Health Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- A4368 - Dose 1 (Experimental): Single dose of A4368 or placebo tablet, orally administered
  Interventions: Drug: A4368 or placebo tablet
- A4368 - Dose 2 (Experimental): Single dose of A4368 or placebo tablet, orally administered
  Interventions: Drug: A4368 or placebo tablet
- A4368 - Dose 3 (Experimental): Single dose of A4368 or placebo tablet, orally administered
  Interventions: Drug: A4368 or placebo tablet
- A4368 - Dose 4 (Experimental): Single dose of A4368 or placebo tablet, orally administered
  Interventions: Drug: A4368 or placebo tablet
- A4368 - Dose 5 (Experimental): Single dose of A4368 or placebo tablet, orally administered
  Interventions: Drug: A4368 or placebo tablet
- A4368 - Dose 6 (Experimental): Single dose of A4368 or placebo tablet, orally administered
  Interventions: Drug: A4368 or placebo tablet
- A4368 - Dose 1 repeated (Experimental): Multiple dose of A4368 or placebo tablet, orally administered daily for 14 consecutive days
  Interventions: Drug: A4368 or placebo tablet
- A4368 - Dose 2 repeated (Experimental): Multiple dose of A4368 or placebo tablet, orally administered daily for 14 consecutive days
  Interventions: Drug: A4368 or placebo tablet

INTERVENTIONS:
Drug: A4368 or placebo tablet — orally administered

SUMMARY:
A4368 is the autophagy activator that is being developed for the treatment of nonalcoholic steatohepatitis.

The goal of the study is to assess the safety, tolerability, and pharmacokinetics in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects
2. Subject with a body weight of ≥ 55.0 kg and within an ideal body weight ± 20%
3. Consent to follow the contraceptive guidance during the treatment period and for at least 3 months after the last dose of study drug
4. Willing and able to sign the informed consent form

Exclusion Criteria:

1. History of or current clinically significant medical illness
2. History of or current gastrointestinal disease or surgery that can influence in pharmacokinetics of study drug
3. Clinically significant history of hypersensitivity to study drug or any of the excipients of study drug
4. Pregnant or lactating woman
5. Clinically significant abnormal laboratory values for hematology, clinical chemistry, or urinalysis
6. Clinically significant abnormal physical examination, vital signs, or 12-lead ECG
7. Heavy alcohol or caffeine intake or heavy smoker
8. Use of study drug in concurrent interventional study within 180 days prior to the first dose of study drug
9. Use of any drug that may affect drug metabolic enzymes within 30 days prior to the first dose of study drug
10. Donation of whole blood within 60 days or apheresis within 30 days prior to the first dose of study drug
11. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 14 days prior to the first dose of study drug

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Up to 21 days
  The number of subjects with adverse events and abnormal laboratory values

SECONDARY OUTCOMES:
Serum concentration of A4368 | From pre-dose to 48 hours post-dose
  The pharmacokinetics of A4368 in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Seunghoon Han, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- AutophagySciences, Seoul, South Korea